CLINICAL TRIAL: NCT03473548
Title: Feasibility of Unattended Home Polysomnography and Comparison to In-laboratory Polysomnography in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201710103
Record Dates: First submitted 2018-03-13; First posted 2018-03-22 (Actual); Results first posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Childhood OSA
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Single-center, un-blinded, feasibility, methods comparison, and non-inferiority study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Unmonitored Polysomnography (Experimental): All eligible subjects will be asked to conduct an unattended, overnight sleep study performed in their home prior to in-laboratory polysomnography, using a standard Type III portable monitor. The type III portable sleep monitor obtaining greater than or equal to 6 hours of data adequate for polysomnography analysis and determination of an apnea hypopnea index (AHI), average SPO2, and SPO2 nadir.
  Interventions: Device: Portable sleep monitor
- In-laboratory Polysomnography (Active Comparator): All eligible subjects will have in-laboratory polysomnography as is routinely performed in the diagnostic work up for suspected sleep disordered breathing.
  Interventions: Other: In-laboratory Polysomnography

INTERVENTIONS:
Device: Portable sleep monitor — Type III at home portable monitor obtaining greater than or equal to 6 hours of data adequate for polysomnography analysis
  Arms: Unmonitored Polysomnography
Other: In-laboratory Polysomnography — Polysomnography testing will determine the sleep stages, apnea hypopnea index (AHI), blood saturation oxygen nadir (SPO2 nadir), and average blood oxygen saturation. A McGill Oximetry Score will also be calculated for the in-laboratory PSG.
  Arms: In-laboratory Polysomnography

SUMMARY:
The purpose of the study is: 1) To assess the feasibility of unmonitored polysomnography and 2) to compare apnea hypopnea index (AHI), average SPO2, and SPO2 nadir between unmonitored polysomnography and in-laboratory polysomnography in pediatric patients.

DETAILED DESCRIPTION:
The purpose of the study proposed is twofold. First Investigators will test the feasibility of conducting portable sleep monitoring in school aged children using the Clevemed Sleepview (www.clevelmed.com), one of the smallest portable sleep monitors commercially available at 57 grams. Second, Investigators will perform a direct comparison between the results obtained with this portable sleep monitor and those obtained from a standard-of-care in-laboratory attended sleep study performed at the St. Louis Children's Hospital Pediatric Sleep Center. These comparisons will be offered to the participants suspected of having sleep disordered breathing who present to the Washington University Pediatric Otolaryngology Department. Investigators will obtain the medical history and medications and results of the sleep study done at SLCH sleep lab from the medical record for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* 5- to 12-years-old
* Parental informed consent
* Suspected Sleep Disordered Breathing

Exclusion Criteria:

* Developmental delay
* Use of home oxygen
* History of Parasomnia (e.g. narcolepsy, restless leg syndrome, somnambulism)
* History of tracheal surgery
* History of tracheal stenosis
* History of Nocturnal Hypoventilation
* History of Central Sleep Apnea
* Use of a Ventilatory Assist Device (e.g. Non-Invasive Positive Pressure Ventilation)

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2019-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Leonard, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients and their families who present to the Washington University Department of Pediatric Otolaryngology with a suspected diagnosis of sleep disordered breathing was given information regarding the study in the office.
Groups:
- Portable Sleep Monitor: Type III portable monitor obtaining greater than or equal to 6 hours of data adequate for polysomnography analysis and determination of an apnea hypopnea index (AHI), average SPO2, and SPO2 nadir.
  Portable sleep monitor: Type III portable monitor obtaining greater than or equal to 6 hours of data adequate for polysomnography analysis and determination of an apnea hypopnea index (AHI), average SPO2, and SPO2 nadir.
Period: Overall Study
Arm/Group | Portable Sleep Monitor | In-laboratory Polysomnography
Started | 11 | 0
Completed | 8 | 0
Not Completed | 3 | 0
Not completed — Did not attempt HST testing | 3 | 0

BASELINE CHARACTERISTICS:
Population: Subjects were identified from patients presenting to the Washington University in St. Louis Pediatric Otolaryngology Clinic who are suspected of having sleep disordered breathing. All 10/11 participants completed an in lab polysomnography.
Groups:
- In Lab Polysomnography: All eligible subjects will have in-laboratory polysomnography as is routinely performed in the diagnostic work up for suspected sleep disordered breathing. The in-laboratory sleep study will be done at the St. Louis Children's Hospital Pediatric Sleep Center, which is an American Academy of Sleep Medicine accredited sleep disorder center. The Center is sound-proof, and has been designed to provide as natural and home-like an atmosphere as possible. Infrared monitoring equipment allows for patient observation from outside of the patient's sleep room. At least one parent is required to stay in the room overnight with the patient. A second parent can stay as well, but not required. The Center is located inside of St. Louis Children's Hospital within an inpatient medical unit, which is staffed with physicians and nurses 24 hours per day
Arm/Group | In Lab Polysomnography
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Standard Deviation); unit: years] — Population: One 1 out of 10 participants had > 6 hours of HST recording and > 6 hours of in lab polysomnography
  years | 7 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Greater Than or Equal to 6 Hours of Sleep Data
Description: Feasibility of obtaining greater than or equal to 6 hours of data adequate for polysomnography analysis and determination of an apnea hypopnea index using un-attended polysomnography; polysomnography analysis will be performed to determine if an apnea hypopnea index can be determined; <5=Normal (no Sleep Apnea); 5-15=Mild Sleep Apnea; 15-30=Moderate Sleep Apnea; >30 Severe Sleep Apnea
Time Frame: greater than or equal to 6 hours
Population: Only 1/10 participant had > 6 hours of collected data on the Home Polysomnography
Measure: Count of Participants; unit: Participants
Arm/Group | Portable Sleep Monitor
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Apnea Hypopnea Index (AHI) Score
Description: Number of participants with Apnea Hypopnea Index (AHI) score
Time Frame: greater than or equal to 6 hours
Population: Only 1/10 participant had > 6 hours of collected data on the Home Polysomnography
Measure: Count of Participants; unit: Participants
Arm/Group | Portable Sleep Monitor
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: SPO2 Result
Description: Number of Participants with an SPO2 result
Time Frame: greater than or equal to 6 hours
Population: Only 1/10 participant had > 6 hours of collected data on the Home Polysomnography
Measure: Count of Participants; unit: Participants
Arm/Group | Portable Sleep Monitor
Number analyzed (Participants) | 1
Participants | 1

4. Secondary Outcome: SPO2 Nadir
Description: Number of participants with an SPO2 nadir
Time Frame: greater than or equal to 6 hours
Population: Only 1/10 participant had > 6 hours of collected data on the Home Polysomnography
Measure: Count of Participants; unit: Participants
Arm/Group | Portable Sleep Monitor
Number analyzed (Participants) | 1
Participants | 1

5. Secondary Outcome: McGill Oximetry Score
Description: Number of participants with McGill Oximetry Score
Time Frame: greater than or equal to 6 hours
Population: Only 1/10 participant had > 6 hours of collected data on the Home Polysomnography
Measure: Count of Participants; unit: Participants
Arm/Group | Portable Sleep Monitor
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was only collected during the HST testing and the in lab PSG testing through study completion, an average of 6 hours.
Description: The investigator will closely monitor subjects for evidence of adverse events. All adverse events will be reported and followed until satisfactory resolution. The description of the adverse experience will include the time of onset, duration, intensity, etiology, relationship to the study (none, unlikely, possible, probable, highly probable), and any treatment required. No Adverse Events meeting the stated definitions occurred.
Arm/Group | Portable Sleep Monitor
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT03473548/Prot_001.pdf